CLINICAL TRIAL: NCT01557140
Title: A Randomized Trial of Carvedilol After Renin-angiotensin System Inhibition in Chronic Chagas Cardiomyopathy
Brief Title: A Randomized Trial of Carvedilol in Chronic Chagas Cardiomyopathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Antonio Luiz Pinho Ribeiro, Director-General, Hospital das Clínicas, UFMG, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Carvedilol in Chagas disease
Record Dates: First submitted 2012-02-21; First posted 2012-03-19 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Chagas Cardiomyopathy; Heart Failure; Dilated Cardiomyopathy
Keywords: Chagas cardiomyopathy,; Renin-angiotensin system,; Beta-blockers,; Enalapril,; Carvedilol,; Renin-angiotensin system inhibitors,; Brain natriuretic peptide level,; Left ventricular ejection fraction,; Chemokines
MeSH Terms: conditions — Chagas Cardiomyopathy; Heart Failure; Cardiomyopathy, Dilated | interventions — Carvedilol; Random Allocation; Double-Blind Method; Control Groups; Clinical Trials as Topic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RASi plus placebo (Placebo Comparator): RAS inhibition was optimized and after patients were randomly assigned to receive placebo
- RASi plus carvedilol (Experimental): RAS inhibition was optimized and after patients were randomly assigned to receive carvedilol
  Interventions: Drug: RASi plus carvedilol

INTERVENTIONS:
Drug: RASi plus carvedilol — Patients were randomly assigned to 2 groups, with 1 group receiving renin-angiotensin system inhibitors (enalapril) plus carvedilol and the other receiving renin-angiotensin system inhibitors (enalapril) plus placebo
  Other Names: Randomized; Double blind; Controlled; Trial
  Arms: RASi plus carvedilol

SUMMARY:
Chronic Chagas cardiomyopathy causes substantial morbidity and mortality in Latin America. Whether RAS inhibitors and beta-blockers are safe and beneficial has been challenged because of the lack of formal trials. Hence, the objective of this study was to determine the safety and efficacy of renin-angiotensin system (RAS) inhibitors and beta-blockers in chronic Chagas cardiomyopathy. This way, the investigators conducted a double-blind, placebo-controlled, and randomized trial in 42 patients with Trypanosoma cruzi infection and cardiomyopathy. All patients received enalapril (up-titrated to 20 mg BID) and spironolactone (25 mg QD). Subsequently, the patients were randomly assigned to receive placebo (n = 20) or carvedilol up-titrated to 25 mg BID (n = 19). The primary end points were change in left ventricular ejection fraction (LVEF) after RAS inhibition and that after the addition of carvedilol. The secondary end points were changes in other echocardiographic parameters, Framingham score, quality of life (36-item Short-Form Health Survey), New York Heart Association class, radiographic indices, brain natriuretic peptide levels, and chemokines as well as safety end points.

DETAILED DESCRIPTION:
Chronic Chagas cardiomyopathy (CCC) is an important cause of heart failure (HF) and sudden death in Latin America.1 According to recent estimates, 13 million people worldwide are infected with Trypanosoma cruzi, of whom 3.0 to 3.3 million are symptomatic.2 The incidence rate is 200000 cases per year. Among those infected, 30% have clinical features of CCC and 15% ultimately develop overt left ventricular (LV) insufficiency-the main prognostic determinant of the disease. In Chagas cardiomyopathy, the hemodynamic and neurohormonal responses do not differ from those in other cardiomyopathies. This common pathophysiology suggests that treatments shown to be effective by classic HF trials should be beneficial in CCC. However, CCC has several specific characteristics, such as early cardiac denervation, frequent ventricular arrhythmias, and several forms as well as grades of conduction disturbances, including sinus bradycardia, complete atrioventricular block, and right bundle-branch block. Morphologically, hypertrophy, dilatation, and severe fibrosis are prominent. In 20% to 40% of cases, an apical ventricular aneurysm is present.1 These peculiarities in combination lead to a high incidence of sudden death (60% of all deaths), cardiac insufficiency, and ventricular remodeling. The responses of patients to the usual drugs prescribed in HF could be different, and this perception has led to the suboptimal dosing or lack of initiation of medical treatments that are of proven efficacy in patients with other etiologies of HF. The underlying problem is that therapies that are effective in patients with HF caused by non-chagasic cardiomyopathies, such as those with renin-angiotensin system inhibitors (RASis) and h-blockers, have yet to be formally tested in CCC. There are few clinical trials and no randomized study on this subject. Consequently, the investigators evaluated the effects of optimizing treatment with enalapril and spironolactone and then undertook a randomized trial of adding a h-blocker in the treatment of patients with CCC.

ELIGIBILITY:
Inclusion Criteria:

* Criteria for inclusion were positivity for T cruzi as confirmed by 2 or more serological tests (indirect immunofluorescence, ELISA, and/or indirect hemagglutination) and having cardiomyopathy.
* Cardiomyopathy was present when at least 3 of the following criteria were fulfilled:

  * LV enddiastolic diameter (LVDD) N55 mm
  * LVDD/body surface area > 2.7cm/m2
  * LV ejection fraction (LVEF) < 55%
  * QRS interval > 120 ms
  * echocardiographic evidence of diffuse or segmental systolic wall motion abnormalities.

Exclusion Criteria:

* Exclusion criteria were being pregnant
* Using any h-blocker
* Having additional comorbidities (eg, hypertension, diabetes mellitus, thyroid dysfunction, chronic obstructive pulmonary disease, asthma, and renal or hepatic failure).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2003-05; Primary Completion 2004-03 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Changes in left ventricular ejection fraction | Baseline, 4 months and 8 months

SECONDARY OUTCOMES:
Changes in Framingham score | Baseline, 4 months and 8 months
Changes in quality of life (36-item Short-Form Health Survey) | Baseline, 4 months and 8 months
Changes in New York Heart Association functional class | Baseline, 4 months and 8 months
Changes in cardiothoracic ratio | Baseline, 4 months and 8 months
Changes in echocardiographic diastolic function indices | Baseline, 4 months and 8 months
Changes in brain natriuretic peptide levels | Baseline, 4 months and 8 months
Changes in chemokines | Baseline, 4 months and 8 months
Changes in autoantibodies levels | Baseline, 4 months and 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Fernando A Botoni, MD, PhD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Chagas Disease Outpatient Center of the Federal University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Result] Botoni FA, Poole-Wilson PA, Ribeiro AL, Okonko DO, Oliveira BM, Pinto AS, Teixeira MM, Teixeira AL Jr, Reis AM, Dantas JB, Ferreira CS, Tavares WC Jr, Rocha MO. A randomized trial of carvedilol after renin-angiotensin system inhibition in chronic Chagas cardiomyopathy. Am Heart J. 2007 Apr;153(4):544.e1-8. doi: 10.1016/j.ahj.2006.12.017. PMID 17383291